CLINICAL TRIAL: NCT00759837
Title: An Open-Label, Single-Dose, Parallel-Group Study of the Pharmacokinetics and Safety of Bosutinib in Subjects With Chronic Hepatic Impairment and in Matched Healthy Adults
Brief Title: Study Evaluating The Pharmacokinetics (PK) And Safety Of Bosutinib In Subjects With Liver Disease And In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 3160A4-1111
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2009-07-16 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer; Leukemia, Myeloid, Chronic
MeSH Terms: conditions — Breast Neoplasms; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of bosutinib and the safety and tolerability of bosutinib in healthy subjects and subjects with liver disease.

ELIGIBILITY:
Inclusion criteria (for both study populations):

1. Men or women of nonchildbearing potential (WONCBP) aged 18 to 65 years inclusive at screening.

   WONCBP may be included if they are either surgically sterile (hysterectomy and/or oophorectomy) or postmenopausal for more than 1 year (with follicle-stimulating hormone [FSH] level greater than or equal to 8 mIU/mL) and must have a negative serum pregnancy test result within 48 hours before administration of test article. Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound scan. Sexually active men must agree to use a medically acceptable form of contraception during the study and continue using it for 12 weeks after test article administration.
2. Have a high probability for compliance with and completion of the study.

Exclusion criteria (for both study populations):

1. History of clinically important cardiovascular disease.
2. Family history of QT prolongation, syncope, seizure, or unexplained cardiac-related death.
3. Presence or history of any disorder that may prevent the successful completion of the study.

Other inclusion and exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Blood samples | 5 weeks

SECONDARY OUTCOMES:
Safety based on adverse events monitoring, physical examinations, vital sign evaluations, 12-lead ECGs and routine laboratory tests. | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Warsaw, Poland